CLINICAL TRIAL: NCT01855542
Title: The Aim of This Investigation is to Compare the Influence of 0.9% Saline and Plasmalyte Solution on Acid-base Balance and Electrolytes in Healthy Patients Undergoing Major Spine Surgeries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4-2012-0059
Record Dates: First submitted 2013-05-07; First posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Spinal Surgery
Keywords: metabolic acidosis, plasmalyte solution, 0.9% normal saline
MeSH Terms: conditions — Acidosis | interventions — Saline Solution; Plasmalyte A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.9% saline (Experimental): In each group, patients received either 0.9% normal saline or plasmalyte solution until end of surgery.
  Interventions: Other: 0.9% normal saline
- plasmalyte (Active Comparator): In each group, patients received either 0.9% normal saline or plasmalyte solution until end of surgery.
  Interventions: Other: plasmalyte

INTERVENTIONS:
Other: 0.9% normal saline — In each group, patients received either 0.9% normal saline or plasmalyte solution until end of surgery.
  Arms: 0.9% saline
Other: plasmalyte — In each group, patients received either 0.9% normal saline or plasmalyte solution until end of surgery.
  Arms: plasmalyte

SUMMARY:
Chloride-rich isotonic crystalloid solutions have been shown to exert electrolyte imbalance and metabolic acidosis in critically ill patients. The aim of this investigation is to compare the influence of 0.9% saline and plasmalyte solution on acid-base balance and electrolytes in healthy patients undergoing major spine surgeries.

ELIGIBILITY:
Inclusion Criteria:

1.50 patients (aged 20-65) undergoing cervical or lumbar spine surgery who were diagnosed spinal stenosis involving more than tow spinal levels.

Exclusion Criteria:

1. ASA class III or IV
2. pregnancy
3. breast feeding
4. lack of mental weakness(including disabled)
5. using diuretics
6. respiratory insufficiency
7. metabolic acidosis or alkalosis
8. coagulation disorder
9. over hydtration
10. renal failure or serum creatinine > 1.4mg/dl
11. anemia (Hemoglobin 9.0<mg/dl)
12. hypernatremia (Na > 145mEq/L)
13. Hyperkalemia (K>5.5mEq/L)
14. psychological medication or any drugs that influences renal clearance

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
base-excess | Change from baseline in base-excess at postoperative 12 h

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Song JW, Shim JK, Kim NY, Jang J, Kwak YL. The effect of 0.9% saline versus plasmalyte on coagulation in patients undergoing lumbar spinal surgery; a randomized controlled trial. Int J Surg. 2015 Aug;20:128-34. doi: 10.1016/j.ijsu.2015.06.065. Epub 2015 Jun 27. PMID 26123384